CLINICAL TRIAL: NCT03455257
Title: Evaluation of a Cash Transfer Program in Low-Income Families in Guinea-Bissau
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Finance, Guinea-Bissau (Other Government)
Collaborators: International Partnership for Human Development (IPHD) (Unknown); National Institute of Statistics (INE) (Unknown); World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1234
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Per Capita Food Consumption Expenditure; Childhood Growth; Childhood Cognition; Anemia; School Registration and Attendence; Diabetes
MeSH Terms: conditions — Anemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participating families are randomized into one of two groups, an assessment-only controls group or a cash transfer group.
Masking Description: Clarify randomization and masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Families assigned to this arm will be assessment only controls that do not receive the cash transfer.
- Intervention (Experimental): Families assigned to this arm will recieve a cash transfer following an in-depth conversation with the head of household and the signing of a contract stating they understand the purpose of the study.
  Interventions: Behavioral: Cash Transfer

INTERVENTIONS:
Behavioral: Cash Transfer — The heads of households will receive a cash transfer for up to 7 family members in the home every quarter. Head of households will be expected to attend meetings every 4 months at their local community health centers led by Community Health Workers (CHW). Meetings will have 2 components: 1) children under 5 will be measured to identify children at risk of malnutrition and 2) group education sessions. There will also be monthly growth monitoring and education sessions led by CHW for a subgroup of head of households with children identified as risk of malnutrition with rapid referrals to regional tertiary clinics for any children with health problems that cannot be addressed by CHW.
  Arms: Intervention

SUMMARY:
This pilot study will test the effect of a cash transfer program aiming to improve family food consumption patterns, family health and schooling, with resulting benefits for childhood growth and cognition.

DETAILED DESCRIPTION:
Cash transfer (CT) programs in low-income countries that allow recipients to receive cash designated for specific household expenditures such as food and family health and education typically show significant program benefits. In particular, several programs have shown positive impacts on use of health care resources, nutrition status and self-reported health, along with significant improvements in the motor and cognitive development of young children.

Guinea-Bissau is currently the 11th poorest country and is thus an appropriate target for a cash transfer program. This project will pilot test the effect of a 2 year cash transfer program aiming to improve family food consumption patterns, family health and schooling, with resulting benefits for childhood growth and cognition. Family-wide assessment will be conducted to examine the impact in all family members. Baseline and 3 follow up assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Families (defined as groups of individuals who routinely eat together) in 3 regions of Guinea-Bissau.
* Identified by developing scale based upon household characteristics and assets per capita. As well as access to services such as water, electricity and sanitation.
* Families having the lowest score identified as lowest income were recruited.

Exclusion Criteria:

* Families with high scores on asset scale.
* Families uninterested in participating.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34148 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in per capita food expeditures | Baseline, year 1, year 2 and year 3
  change in per capita food expenditure per family will be calculated.

SECONDARY OUTCOMES:
Changes in family demographics | Baseline, year 1, year 2 and year 3
  Changes in family demographics will be tracked.
Change in weight | Baseline, year 1, year 2 and year 3
  Change in weight for all participants in the study and children born after cash transfer program starts.
Change in height | Baseline, year 1, year 2 and year 3
  Change in height for all participants in the study and children born after cash transfer program starts.
Change in mid-upper arm circumference (MUAC) | Baseline, year 1, year 2 and year 3
  Change in MUAC for all participants in the study and children born after cash transfer program starts.
Change in waist circumference | Baseline, year 1, year 2 and year 3
  Change in waist circumference for all participants in the study and children born after cash transfer program starts.
Change in hemoglobin | Baseline, year 1, year 2 and year 3
  Change in hemoglobin for pregnant women, children born after the program begins, older children born in 2003, 2010, 2014.
Change in blood pressure | Baseline, year 1, year 2 and year 3
  Change in blood pressure will be measured in 100 randomly selected families in each region with a family size 2-4 and 5-8.
Change in HbA1c | Baseline, year 1, year 2 and year 3
  Change in HbA1c will be measured in 100 randomly selected families in each region with a family size 2-4 and 5-8.
Food intake | Year 1, year 2 and year 3
  Food intake assessment
Cognition function | When children are 18th months
  Children born after the cash transfer progam will have a single cognitive function test at 18 months of age.
Change in school attendence | Each semester of school in year 1, 2 and 3 of study
  School enrollment, attendance, drop out and grade graduation will be assessed for all children through data extraction from school records.
Change in head circumference | After birth, year 1, year 2, year 3
  Children born after the cash transfer progam will have head circumference taken.
Change in Literacy | Year 1, year 2, year 3
  Children 7 and 14 will complete literacy testing.
Change in Grip Strength | Baseline, year 1, year 2 and year 3
  Change in grip strength will be measured in 100 randomly selected families in each region with a family size 2-4 and 5-8.

CONTACTS AND LOCATIONS:
Overall Officials: Alfa U Jalo, MS, Principal Investigator — Ministry of Finance
Locations (1):
- PDDC, Bissau, Guinea-Bissau